CLINICAL TRIAL: NCT00048321
Title: ISIS 104838-CS7, A Double-Blind, Placebo-Controlled, Randomized Trial of the Safety, Efficacy and Pharmacokinetic Profile of ISIS 104838 (TNF-alpha Antisense Oligonucleotide) Subcutaneous Injections in Active Rheumatoid Arthritis Patients
Brief Title: ISIS 104838, an Inhibitor of Tumor Necrosis Factor, for Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 104838-CS7
Record Dates: First submitted 2002-10-29; First posted 2002-10-31 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2007-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ISIS104838

INTERVENTIONS:
Drug: ISIS 104838

SUMMARY:
ISIS 104838 is an antisense oligonucleotide drug that reduces the production of a specific protein called tumor necrosis factor (TNF-alpha), a substance that contributes to joint pain and swelling in rheumatoid arthritis. ISIS 104838 works by blocking TNF-alpha messenger RNA, the "instruction" molecule that is required for the production of TNF-alpha protein. This trial will assess the safety and efficacy of ISIS 1048383 by subcutaneous injection, administered by 3 different dosing regimens for 3 months, versus placebo. Approximately 160 TNF-alpha inhibitor-naïve rheumatoid arthritis patients will be evaluated at 32 sites in the U.S. and Canada.

ELIGIBILITY:
Inclusion Criteria

1. Age >/= 18 years.
2. Rheumatoid arthritis for >/= 6 months.
3. Active disease as defined by >/= 6 swollen and >/= 9 tender joints, AND an abnormal C-reactive protein or Westergren Erythrocyte Sedimentation Rate lab test, OR Morning Stiffness >/= 1 hour.
4. Use of at least one DMARD, and ability to discontinue any current DMARD.

Exclusion Criteria

1. Onset of rheumatoid arthritis before the 16th birthday.
2. Wheelchair or bed-bound functional level.
3. No previous infliximab or etanercept treatment, or investigational therapy (not placebo) with other TNF-alpha inhibitors.
4. Prednisone > 10 mg per day or more than one nonsteroidal anti-inflammatory drug.
5. Patients with an active infection, a history of tuberculosis, multiple sclerosis, other poorly controlled medical illness, or a malignancy within the last 5 years.
6. Patients who require intravenous heparin therapy or with a history of a bleeding problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-01-01 (Actual); Primary Completion 2003-02-01 (Actual); Study Completion 2003-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (26):
  - Birmingham, Alabama
  - Paradise Valley, Arizona
  - Los Angeles, California
  - Rancho Cucamonga, California
  - Fort Lauderdale, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Wichita, Kansas
  - Louisville, Kentucky
  - Greenbelt, Maryland
  - Fall River, Massachusetts
  - Lansing, Michigan
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Mayfield, Ohio
  - Duncansville, Pennsylvania
  - Willow Grove, Pennsylvania
  - Amarillo, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Lubbock, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Canada (5):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario

REFERENCES:
- [Derived] Burel SA, Machemer T, Baker BF, Kwoh TJ, Paz S, Younis H, Henry SP. Early-Stage Identification and Avoidance of Antisense Oligonucleotides Causing Species-Specific Inflammatory Responses in Human Volunteer Peripheral Blood Mononuclear Cells. Nucleic Acid Ther. 2022 Dec;32(6):457-472. doi: 10.1089/nat.2022.0033. Epub 2022 Aug 17. PMID 35976085
- See also: Type "ISIS 104838" in search box — http://www.centerwatch.com